CLINICAL TRIAL: NCT03376672
Title: A Prospective Phase 2 Study to Assess the Minimal Residual Disease After Ixazomib Plus Lenalidomide Plus Dexamethasone (IRd) Treatment for Newly Diagnosed Transplant Eligible Myeloma Patients
Brief Title: Ixazomib Plus Lenalidomide Plus Dexamethasone for Newly Diagnosed Myeloma Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Raija Silvennoinen (Other)
Collaborators: Nordic Myeloma Study Group (Other); Celgene (Industry); Takeda (Industry)
Responsible Party: Sponsor-Investigator, Raija Silvennoinen, Principal Investigator, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMSG#23/15
Record Dates: First submitted 2017-12-03; First posted 2017-12-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ixazomib,lenalidomide,dexamethasone (Experimental): Ixazomib capsules 4Mg Oral capsule on days 1, 8 and 15 in 28d cycle, lenalidomide 25 milligram capsules on days 1-21 in 28d cycle, dexamethasone 40 milligram capsules on days 1, 8, 15, 22 in 28d cycle
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone
- High risk maintenance arm (Experimental): Ixazomib capsules 4Mg Oral capsule on days 1, 8, 15, lenalidomide 10 milligram on days 1-21 in 28d cycle
  Interventions: Drug: Ixazomib; Drug: Lenalidomide
- Standard and low risk maintenance arm (Experimental): Lenalidomide
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Ixazomib — All patients will have similar induction and consolidation treatment with the same regimen.
  Arms: High risk maintenance arm; Ixazomib,lenalidomide,dexamethasone
Drug: Lenalidomide — All patients will have similar induction and consolidation treatment with the same regimen.
Drug: Dexamethasone — All patients will have similar induction and consolidation treatment with the same regimen.
  Arms: Ixazomib,lenalidomide,dexamethasone

SUMMARY:
This study will evaluate the efficacy and safety of 3-drug all-oral combination, ixazomib plus lenalidomide plus dexamethasone (IRd) as induction treatment for autologous stem cell transplantation eligible patients followed by IRd consolidation and risk based maintenance treatment with IR or R alone.

DETAILED DESCRIPTION:
This Nordic Myeloma Study Group study is phase 2 study for newly diagnosed transplant eligible myeloma patients between 18 - 70 years of age. Patients will have four IRd cycles of 28 day each as induction consisting of ixazomib 4 mg on days 1, 8 and 15 and lenalidomide 25 mg on days 1-21 and dexamethasone 40 mg on days 1, 8, 15 and 22. After autologous stem cell mobilisation and transplantation patients will receive 2 consolidation cycles with the same combination as during induction. This is followed by risk based maintenance so that high-risk patients will have ixazomib plus lenalidomide maintenance and standard-low risk patients lenalidomide alone. The treatment will continue until progression or excess toxicity. The primary endpoint is minimal residual disease < 0.01% assessed by 8-color flow cytometry (EuroFlow) and secondary endpoint is achievement of minimal residual negativity status assessed by 8-color flow cytometry. Other secondary endpoints are safety, improvement of response during maintenance treatment, progression free survival, time to next treatment, quality of life and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed transplant eligible male or female multiple myeloma patients, 18-70 years of age, who have not received prior treatment for multiple myeloma
2. Symptomatic and measurable disease diagnosed by standard criteria (International Myeloma Working Group, CRAB criteria)
3. Voluntary written informed consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
4. Female patients who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, fertile, agree to practice 2 effective methods of contraception, at the same time, and agree to ongoing pregnancy testing and adhere to the guidelines of the lenalidomide pregnancy prevention program from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

• Agree to practice effective barrier contraception and adhere to the guidelines of the lenalidomide pregnancy prevention program during the entire study treatment period and through 90 days after the last dose of study drug, OR

* Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.

  4. Patients must have a diagnosis of a symptomatic multiple myeloma without any previous therapies except dexamethasone 160 mg dose, or comparable dose of other steroids, and local radiotherapy for symptom control 5. Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2.

  6. Patients must meet the following clinical laboratory criteria:
* Absolute neutrophil count (ANC) ≥ 1,000/mm3 (≥ 1.0 x 109/L) and platelet count ≥ 75,000/mm3 (75 x 109/L). Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
* Total bilirubin ≤ 1.5 × the upper limit of the normal range (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN.
* Calculated creatinine clearance ≥ 30 mL/min (Cockcroft-Gault estimation of creatinine clearance (CRcl): CRcl (mL/min) = (140 - age) (weight [kg]) / 72 (serum creatinine [mg/dL]); for females, multiply by 0.85 (Cockcroft DW. 1976, Luke DR. 1990).

  7. Patient must be willing and able to adhere to the study protocol visit schedule and other protocol requirements.

  8. Negative pregnancy test at inclusion if applicable

Exclusion Criteria:

* 1. Female patients who are lactating or have a positive serum pregnancy test during the screening period.

  2. Major surgery within 14 days before enrollment. 3. Radiotherapy within 14 days before enrollment 4. Central nervous system involvement with multiple myeloma. 5. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.

  6. Inability, unwillingness or contraindication to use thrombosis prophylaxis or antithrombotic therapy or herpes zoster prophylaxis 7. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.

  8. Systemic treatment, within 14 days before the first dose of ixazomib, strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.

  9. Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.

  10. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.

  11. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.

  12. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib or lenalidomide including difficulty swallowing.

  13. Diagnosed or treated for another malignancy within 5 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

  14. Patient has Grade 1 polyneuropathy with pain on clinical examination during the screening period.

  15. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.

  16. Patients that have previously been treated for multiple myeloma or smoldering myeloma with ixazomib or any other therapy, or participated in a study with ixazomib whether treated with ixazomib or not.

  17. Primary plasma cell leukemia, POEMS syndrome, Waldenström disease, myelodysplastic syndrome or myeloproliferative disease

  18. Systemic AL amyloidosis/primary amyloidosis or myeloma associated amyloidosis.

  19. Allogeneic stem cell transplantation planned

  20. Participants receiving any other investigational agents or received within 60 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Flow cytometric assessment < 0.01% | 48 months
  Minimal residual disease by multiparameter flow cytometry (MFC) < 0.01%

SECONDARY OUTCOMES:
Flow cytometry negativity | 48 months
  Minimal residual disease negativity by MFC

OTHER OUTCOMES:
Overall survival | Up to 10 years
  Survival time
Progression free survival | Up to 10 years
  Time without progression of myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Raija H Silvennoinen, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (26):
- Finland (9):
  - Helsinki University Central Hospital, Helsinki
  - Central Finland Central Hospital, Jyväskylä
  - Kainuu Central Hospital, Kajaani
  - Kymenlaakso Central Hospital, Kotka
  - Kuopio University Hospital, Kuopio
  - Päijät-Häme Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- VIlnius University Hospital, Vilnius, Lithuania
- Norway (4):
  - Forde Central Hospital South, Førde
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - Trondheim University Hospital, Trondheim
- Sweden (12):
  - Borås University Hospital, Borås
  - Göteborg University Hospital, Gothenburg
  - Halmstad Hospital Region Halland, Halmstad
  - Linköping University Hospital, Linköping
  - Sunderby Hospital Region Norrbotten, Luleå
  - Lund University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Helsingborg Hospital Skane, Skåne
  - Karolinska University Hospital, Stockholm
  - Uddevalla Hospital, Uddevalla
  - Uppsala University Hospital, Uppsala
  - Varberg Hospital, Varberg

IPD SHARING:
Plan to Share IPD: No